CLINICAL TRIAL: NCT01725464
Title: The Effect of Nasal Cannula During the First 2 Hours Postoperative in Patient Undergoing Thoracotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Profesor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 541/2555(EC)
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Lung Surgery; Hypoxia; Postoperative
Keywords: thoracotomy; oxygen saturation; postoperative
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oxygen cannular (Experimental): Patient receives oxygen supplementation 5 LPM via oxygen cannular for 120 minutes after the operative
  Interventions: Device: oxygen cannular

INTERVENTIONS:
Device: oxygen cannular — Patient receives oxygen supplementation 5 LPM via oxygen cannular for 120 minutes after the operative

SUMMARY:
During early postoperative after lung resection surgery, patients without oxygen supplementation may experience hypoxemia. Oxygen supplementation can be given via oxygen mask or cannular. In this study the investigators want to the sudy the effect of oxygen supplementation via oxygen cannular during the first 120 minutes after surgery

ELIGIBILITY:
Inclusion Criteria:

* age =/> 18 years
* lobectomy or pneumonectomy or wedge resection
* ASA 1-3
* preoperative oxygen saturation < 95 %
* receiving epidural analgesia

Exclusion Criteria:

- cannot communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mean oxygen saturation at 30 minutes postoperative | 30 minutes

SECONDARY OUTCOMES:
incidence of oxygen saturation < 95% between 120 minutes until 3 days postoperative | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Sirilak Suksompong, Bangkok, Thailand